CLINICAL TRIAL: NCT02472834
Title: Amino Acid Therapy to Modify Protein Carbamylation in End Stage Renal Disease: A Randomized Trial
Brief Title: Trial of Carbamylation in Renal Disease-Modulation With Amino Acid Therapy
Acronym: CarRAAT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sahir Kalim, Assistant Professor in Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-P-000562; 5K23DK106479-04 (NIH)
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Carbamylation; Albumin; Protein structure; Kidney disease
MeSH Terms: conditions — Kidney Diseases | interventions — Amino Acids, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amino acid supplementation NephrAmine® (Experimental): 250 mL of 5.4% amino acid solution (NephrAmine) by intravenous infusion 3 x weekly for 8 weeks plus 4 weeks of follow-up.
  Interventions: Dietary Supplement: Amino acid supplementation NephrAmine®
- Standard-of-care (No Intervention): Standard-of-care does not include amino acid supplementation, but this control arm will be evaluated for the same outcomes as the experimental arm for 8 weeks plus 4 weeks of follow-up

INTERVENTIONS:
Dietary Supplement: Amino acid supplementation NephrAmine® — Dialysis patients will be randomized to receive either 250 mL of NephrAmine® (5.4% amino acids for injection; B. Braun Medical, Inc) containing ~14 grams of essential amino acids during each dialysis session (3 times weekly for 8 weeks) or no treatment (standard-of-care)
  Other Names: NephrAmine®
  Arms: Amino acid supplementation NephrAmine®

SUMMARY:
Patients with end stage renal disease (ESRD) usually have high levels of urea that may interact with blood proteins and change their structure by a process known as carbamylation. Evidence suggests that high levels of carbamylated proteins may be linked to adverse outcomes in dialysis patients. This is a randomized, open-label study to evaluate the effects of amino acid supplementation on levels of carbamylated proteins in ESRD patients. Secondary objectives will be to determine whether this intervention can modify intermediate markers of inflammation, cardiac stress, and erythropoietin responsiveness in this population. Sixty ESRD patients on dialysis will be randomized into two groups of 30 patients each. Group 1 will receive intravenous supplementation with an FDA-approved amino acid solution (250 mL of NephrAmine®, 5.4% amino acids) during regular dialysis sessions (3 times weekly for 8 weeks); Group 2 will be treated according to standard-of-care (no amino acid supplementation). During the 8 weeks of therapy and for 4 weeks of follow-up, blood will be drawn from patients' existing hemodialysis access ports (~20 mL once per month) to measure levels of carbamylated albumin, amino acids, selected biomarkers, and standard laboratory values. Patients randomized to Group 1 will have fluid volume equivalent to the amino acid therapy removed by ultra-filtration to avoid net fluid gain. All patients will be monitored for safety (adverse events) and for changes in hemodynamics and dialysis prescription.

DETAILED DESCRIPTION:
As human kidney function declines, so does the kidney's ability to excrete urea, the chief end product of nitrogen metabolism. Excess urea may accelerate the pathophysiological consequences of kidney failure. Urea spontaneously dissociates to form cyanate, which, in its unprotonated form can react with protein amino groups in a process known as carbamylation. Carbamylation-induced protein alterations may be involved in the progression of various diseases by changing the structure, charge, and function of enzymes, hormones, receptors, and amino acids. For example, proteins such as collagen and low density lipoproteins (LDLs), when carbamylated, have been shown to induce the characteristic biochemical events of atherosclerosis progression. This research aims to evaluate whether amino acid supplementation can attenuate such processes that are known to contribute to morbidity in patients with ESRD.

Percent carbamylated albumin (C-Alb) level will be used as a measure of overall carbamylation burden. Previous studies conducted by MGH Investigators have shown a negative correlation between %C-Alb and circulating amino acids, suggesting that free amino acids may actively scavenge reactive isocyanate. Further, ex vivo studies show that amino acid supplementation reduces the carbamylation reaction. The MGH Investigators recently demonstrated an association between markers of cardiac stress, heart failure and carbamylation in patients with ESRD and found that %C-Alb was strongly associated with erythropoietin resistance in dialysis patients. Additionally, using validated measures of total-body carbamylation, these and other Investigators have reported that elevated protein carbamylation was linked with higher mortality in several distinct ESRD cohorts. Finally, preliminary data from a recent pilot study at MGH (NCT01612429) suggests that amino acid supplementation in patients with ESRD undergoing maintenance hemodialysis can attenuate carbamylation of proteins.

The proposed randomized study will directly evaluate the impact of amino acid supplementation on: (1) the burden of carbamylation in terms of %C-Alb; and (2) selected intermediate determinants of clinical outcomes, i.e., markers of inflammation, cardiac stress, and erythropoietin responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the investigational nature of the study and sign written informed consent
* Willing and able to adhere to all study-related procedures, including adherence to study medication regimen
* ≥18 years old
* On stable medical therapy in the last 30 days before the study entry, defined as no change, addition, or removal of medications
* Patients must satisfy the following criteria based on the initial screening laboratory values:

  * Serum albumin ≥ 3.0 g/dL (30 g/L)
  * Dialysis adequacy recorded as Kt/ V > 1.2
  * Carbamylated albumin (C-Alb) > 7.7 mmol/mol
* Women of childbearing potential must be practicing barrier or oral contraception, for the duration of the study-related treatment, or be documented as surgically sterile or one year post-menopausal
* If female, be non-nursing, non-pregnant and have a negative pregnancy test within two weeks of starting study treatment
* On stable hemodialysis therapy for at least 90 days before the study entry, defined as receiving thrice weekly dialysis and carrying a diagnosis of ESRD
* Prescribed a dialysis treatment time of 4 hours per session

Exclusion Criteria:

* Taking any type of amino acid supplementation within the last 90 days
* Received parenteral nutrition within last 90 days
* History of allergy to any amino acid compound
* Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg during any of the previous 3 dialysis sessions (confirmed by repeat)
* Severe hepatic impairment
* HIV positive
* Condition with prognosis <1 year at time of study entry
* Body Mass Index (BMI) <18 or >30
* Current active treatment in another investigational study or participation in another investigational study in the 1 month prior to screening
* Active malignancies or other serious concurrent or recent medical or psychiatric condition which, in the opinion of the Investigator, makes the patient unsuitable for participation in this study
* Presence of asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Differences in plasma carbamylated albumin (C-Alb) levels | Baseline and weeks 4, 8, and 12

SECONDARY OUTCOMES:
Safety of amino acid infusion | Baseline and weeks 4, 8, and 12
  In terms of in terms of adverse events, changes in amino acid levels, ammonia, routine dialysis labs, intra-dialytic hemodynamics, and dialysis prescription during 8 weeks of therapy and 4 weeks of follow-up post-therapy
Differences in cardiac markers | Baseline and weeks 4, 8, and 12
  Changes in Troponin T and NT-Pro-BNP during 8 weeks of therapy and 4 weeks of follow-up post-therapy
Differences in inflammatory markers | Baseline and weeks 4, 8, and 12
  Changes in myeloperoxidase, IL-6, IL-12, IFN-γ, and TNF-α during 8 weeks of therapy and 4 weeks of follow-up post-therapy
Differences in erythropoietin resistance | Baseline and weeks 4, 8, and 12
  Measured in terms of the erythropoietin responsiveness index (ERI, defined as average weekly erythropoietin dose [U]/ kg body weight/ average hemoglobin [g/dL]) (Kalim et al. 2013) during 8 weeks of therapy and 4 weeks of follow-up post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sahir Kalim, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fresenius Medical Centers (local affilliates), Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drechsler C, Kalim S, Wenger JB, Suntharalingam P, Hod T, Thadhani RI, Karumanchi SA, Wanner C, Berg AH. Protein carbamylation is associated with heart failure and mortality in diabetic patients with end-stage renal disease. Kidney Int. 2015 Jun;87(6):1201-8. doi: 10.1038/ki.2014.429. Epub 2015 Feb 11. PMID 25671766
- [Background] Kalim S, Tamez H, Wenger J, Ankers E, Trottier CA, Deferio JJ, Berg AH, Karumanchi SA, Thadhani RI. Carbamylation of serum albumin and erythropoietin resistance in end stage kidney disease. Clin J Am Soc Nephrol. 2013 Nov;8(11):1927-34. doi: 10.2215/CJN.04310413. Epub 2013 Aug 22. PMID 23970130
- [Background] Berg AH, Drechsler C, Wenger J, Buccafusca R, Hod T, Kalim S, Ramma W, Parikh SM, Steen H, Friedman DJ, Danziger J, Wanner C, Thadhani R, Karumanchi SA. Carbamylation of serum albumin as a risk factor for mortality in patients with kidney failure. Sci Transl Med. 2013 Mar 6;5(175):175ra29. doi: 10.1126/scitranslmed.3005218. PMID 23467560
- [Background] Koeth RA, Kalantar-Zadeh K, Wang Z, Fu X, Tang WH, Hazen SL. Protein carbamylation predicts mortality in ESRD. J Am Soc Nephrol. 2013 Apr;24(5):853-61. doi: 10.1681/ASN.2012030254. Epub 2013 Feb 21. PMID 23431074